CLINICAL TRIAL: NCT03570684
Title: Utility of Cable Tie in Laparoscopic Anterior Resection of Rectal Cancer to Decline Reloads of Endoscopic Linear Cutter During the Transection of Rectum
Brief Title: Utility of Cable Tie to Decline Reloads in Laparoscopic Anterior Resection of Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, professor, West China Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRCmodifiedTec01
Record Dates: First submitted 2018-05-05; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Modification of Rectal Cancer Surgery

STUDY DESIGN:
Intervention Model Description: comparing the recent tie used patients with the previous respective data.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tie group (Experimental): During the operation, after mobilization the rectum, the disinfected Cable Tie was introduced into the pelvic cavity.then the rectum was bundled by the tie which was much easier as the tie is auto-locked. pulling the tie and the rectum would be explored clearly, and then the endoscopic linear cutter was introduced to transect the rectum.
  Interventions: Device: Cable Tie
- non-tie group (No Intervention)

INTERVENTIONS:
Device: Cable Tie — During the operation, after mobilization the rectum, the disinfected Cable Tie was introduced into the pelvic cavity.then the rectum was bundled by the tie which was easy as the tie is auto-locked. pulling the tie and the rectum would be explored clearly, and then the endoscopic linear cutter was introduced to transect the rectum. the tie made the rectum folded not applanate, that the cutter was able to transect the rectum easily and with less reloader. when the rectum was resected completely, the tie was get out with the specimen, and do not live in the abdomen.
  Arms: tie group

SUMMARY:
During the laparoscopic anterior resection of rectal cancer, transecting the mobilized rectum in the narrow pelvic was difficult and sometimes need 2-3 reloads of the endoscopic linear cutter. also the angles between the 2-3 staple line threaten the next anastomosis. this study was to explore the Cable Tie to facilitate the transection of rectum and decline the usage of the reloads.

DETAILED DESCRIPTION:
In the modern laparoscopic colorectal surgery, application of endoscopic stapler was necessary and popular, especially in rectal cancer. In the anterior resection of rectal cancer, usage of stapler increase the anal preservation. However during the laparoscopic anterior resection, transecting the mobilized rectum in the narrow pelvic was difficult, even with the flexible linear cutter. 1 reloads of the stapler was unable to transect the rectum completely, and need 2-3 reloads, especially in some fat patients, which was uneconomic.Also increased reloads increase the staple line, and 2 or 3 staple line threaten the next anastomosis, and increasing anastomotic leak rate. this study was to explore the Cable Tie to facilitate the transection of rectum and decline the usage of the reloads. During the operation, after mobilization the rectum, the disinfected Cable Tie was introduced into the pelvic cavity.then the rectum was bundled by the tie which was much easier as the tie is auto-locked. pulling the tie and the rectum would be explored clearly, and then the endoscopic linear cutter was introduced to transect the rectum. the tie made the rectum folded not applanate, that the cutter was able to transect the rectum easily and with less reloader.

ELIGIBILITY:
Inclusion Criteria:

1. rectal cancer patients;
2. the tumor located 5-12cm from the anal verge, that an anterior resection was needed.
3. the cancer has no organ invasion.

Exclusion Criteria:

patients refuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-08-30 (Estimated); Study Completion 2019-03-02 (Estimated)

PRIMARY OUTCOMES:
the number of reloads during the surgery | during the operation
  the number of reloads during the surgery
ratio of patients with 2 or more reloads | during the operation
  ratio of patients with 2 or more reloads

SECONDARY OUTCOMES:
rate of anastomotic leaks | 3 month after the surgery
  rate of anastomotic leaks
operation duration time | during the operation
  operation duration time
complication rate | 3 month after the surgery
  the complication of the operation

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Bi L, Deng X, Meng X, Yang X, Wei M, Wu Q, Ren M, Wang Z. Ligating the rectum with cable tie facilitates rectum transection in laparoscopic anterior resection of rectal cancer. Langenbecks Arch Surg. 2020 Mar;405(2):233-239. doi: 10.1007/s00423-020-01863-6. Epub 2020 Apr 8. PMID 32266529